CLINICAL TRIAL: NCT06754553
Title: Randomized Placebo Controlled Trial Evaluating the Efficacy of Pimavanserin, a Selective Serotonin 5-HydroxyTryptamine-2A (5HT2A) Inverse Agonist, to Treat Impulse Control Disorders in Parkinson's Disease.
Brief Title: Trial Evaluating the Efficacy of Pimavanserin, a Selective Serotonin 5-HydroxyTryptamine-2A (5HT2A) Inverse Agonist, to Treat Impulse Control Disorders in Parkinson's Disease.
Acronym: RETRO-PIMPARK
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Collaborators: NS-PARK Network (Unknown); EUCLID Clinical Trial Platform (Other); F-CRIN (Unknown)
Responsible Party: Sponsor
Other Study IDs: 9552
Record Dates: First submitted 2024-12-30; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Parkinson Disease
Keywords: Pimavanserin; Impulse Control Disorder; Serotoninergic 5-HT2A inverse agonist; Dopamine agonist
MeSH Terms: conditions — Parkinson Disease; Disruptive, Impulse Control, and Conduct Disorders | interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Experimental: PIMAVANSERIN: In this arm, each patient took orally, once daily 2 tablets of active drug pimavanserin of 17mg each during the 8-weeks treatment period.
  Interventions: Behavioral: Assessment of severity of ICD (impulse control disorders); Behavioral: Assessment of motor and non-motors symptoms of PD Evaluation of hyper- and hypodopaminergic behaviors; Behavioral: Assessment of quality of life; Behavioral: Assessment of depression; Behavioral: Assessment of cognition; Behavioral: Assessment of severity of Parkinson Disease; Procedure: Cardiac monitoring
- Placebo: In this arm, each patient took orally, once daily, 2 tablets of matching placebo (containing all of the same excipients except for the active compound) during the 8-weeks treatment period.
  Interventions: Behavioral: Assessment of severity of ICD (impulse control disorders); Behavioral: Assessment of motor and non-motors symptoms of PD Evaluation of hyper- and hypodopaminergic behaviors; Behavioral: Assessment of quality of life; Behavioral: Assessment of depression; Behavioral: Assessment of cognition; Behavioral: Assessment of severity of Parkinson Disease; Procedure: Cardiac monitoring

INTERVENTIONS:
Behavioral: Assessment of severity of ICD (impulse control disorders) — Questionnaire for impulsive-compulsive disorders in Parkinson's disease rating scale (QUIP-RS) administered at day 0, day 28 (Week 4) and day 56 (Week 8)
Behavioral: Assessment of motor and non-motors symptoms of PD Evaluation of hyper- and hypodopaminergic behaviors — Hyper- and hypodopaminergic behaviors (Ardouin's scale); Movement disorders society sponsored unified Parkinson's disease rating scale (MDS-UPDR), and daytime and night time sleep by scale for outcomes in Parkinson's disease SLEEP (SCOPA-SLEEP, ISI, PDSS-2) administered at day 0, day 28 (Week 4) and day 56 (Week 8)
Behavioral: Assessment of quality of life — Parkinson's Disease questionnaire (PDQ-39) administered at day 0, day 28 (Week 4) and day 56 (Week 8)
Behavioral: Assessment of depression — Montgomery-Åsberg Depression Rating Scale (MADRS) administered at day 0 and day 56 (week 8)
Behavioral: Assessment of cognition — Cognitive state of patients by Montreal Cognitive Assessment (MOCA) assessed at day 0
Behavioral: Assessment of severity of Parkinson Disease — Clinical Global Impression Severity scale (CGIS) administered at day 0 , day 7, day 14, day 28, day 42 and day 56 (week 8) and day 112 (Week 16)
Procedure: Cardiac monitoring — Electrocardiogram realized at day 0, 28 and 56.

SUMMARY:
There is no consensus on the treatment of Impulse Control Disorder (ICD) in Parkinson Disease (PD) though it is recommended to reduce the dosage of dopamine agonists (DA).

Reduction of DA frequently leads to a worsening of motor signs (parkinsonism or dyskinesias due to the concomitant increase of levodopa doses) and non-motor signs with the appearance of a DA withdrawal syndrome (DAWS).

Chronic stimulation of the sub-thalamic nuclei may reduce ICD but is restricted to a minority of patients and cases of new-onset ICD symptoms post stimulation have been reported. The benefit of amantadine in pathological gambling is controversial and the efficacy of clozapine has been reported in a few cases but with serious safety limitations. Very recently, naltrexone did not significantly improve ICD.

Thus, an efficacious and safe treatment of ICD in PD remains an unmet need for clinical practice.

Recently, it has been reported that pimavanserin, a selective serotonin 5-HT2A inverse agonist with a satisfactory safety profile without motor side effects, was efficient in improving psychosis, insomnia and day-time sleep in PD.

Pimavanserin, marketed under the tradename NUPLAZID® was approved in 2016 by the U.S. Food and Drug Administration (FDA) for the treatment of hallucinations and delusions associated with Parkinson's disease psychosis.

The link between serotonin and ICD has been well established, since the enhancement of 5HT2A receptors stimulation is associated to ICD, since serotonin modulates mesolimbic dopaminergic reward system transmission and given that serotonin neurotransmission is increased during chronic intake of dopamine agonist such as pramipexole which is well-known to induce ICD in PD patients. Thus, there is a large body of evidence suggesting that the decrease of the 5HT2A activity could be efficient in reducing ICD in PD. This further supports the concept of testing the efficacy of pimavanserin (a selective 5HT2A inverse agonist) for treating ICD in PD. Our aim is to conduct a study evaluating the efficacy and safety of pimavanserin on ICD in PD.

ELIGIBILITY:
Inclusion Criteria:

* Patient with PD according to the UKPDSBB criteria for at least 1 year before randomization
* Patient, man or woman, aged from 35 to 75 years old
* Patient with moderately severe ICD assessed by QUIP-RS (each item being rated 0-16) defined as:

a combined ICD total score (defined as the sum of the 4 ICD sub-scores (pathological gambling + buying + hypersexuality + eating)) superior or equal to 10 or, at least one of the 4 ICD sub-scores in the following range:

"pathological gambling" sub-score from 6 to 12 (included), "buying" sub-score from 8 to 12 (included), "hypersexuality" sub-score from 8 to 12 (included), "eating" sub-score from 7 to 12 (included) (Weintraub et al., 2012). The use of "lower" margins will guarantee that the patient experiences behavioral disturbances severe enough to justify pimavanserin treatment. On the other hand, the use of "upper" margins will guarantee that the patients included in the trial will not suffer from ICD severe enough to question ethically the use of placebo during the 8 weeks of the treatment. Eligibility of patients with QUIP-RS sub-scores above 12 will be assessed upon investigator's request by an adjudication committee composed by independent experts external to the study

* ICD onset after PD onset and after initiation of dopaminergic drugs
* Patient treated by dopaminergic drugs for at least 3 months before randomization in the PIMPARK study
* Patient treated with a stable regimen of levodopa, dopamine agonists, COMT and MAOB inhibitors, amantadine, anticholinergic, antidepressant and benzodiazepine for at least 1 month before the randomization and be willing to remain on the same doses throughout the course of their participation in the trial (Papay et al., 2014)
* Patient with health insurance
* Patient/ guardian / curator who sign the written informed consent for the PIMPARK study
* For women of childbearing potential, use of an effective contraception method for at least 1 month prior to randomization in the PIMPARK study until 8 weeks after the last dose of study drug administration.
* Having participated in the PHRC N 2015 - HUS N°6398 study (PIMPARK study) during the period from 23/10/2020 to 17/06/2024.
* Not objecting, after information, to the reuse of its data from the study PHRC N 2015 - HUS N°6398 for the purposes of this research.

Exclusion Criteria:

* Patient suffering from another parkinsonian syndrome (multiple system atrophy, progressive supranuclear palsy, Lewy body dementia, corticobasal degeneration)
* Patient who have a known hypersensitivity to the study treatment, based on known allergies to drugs of the same class
* Stroke, uncontrolled serious medical illness, myocardial infarction, congestive heart failure, cardiac function disorders, within 6 months before randomization
* Patient with history of long QT syndrome
* Patient with long QTcB detected with ECG at inclusion visit (> 450 ms)
* Patient treated with antipsychotic drugs during the last three months before randomization in the PIMPARK study
* Patient treated with concomitant medication leading to torsade de pointes (TdP) without discontinuation ≥ 5 half-lives before randomization (please refer to medications list with known risks of TdP on appendix XVII.5.10 and check website https://crediblemeds.org/index.php/tools/ for the most up-to-date information)
* Patient with hydro-electrolytics troubles, particularly hypokaliemia or hypocalcemia not corrected, at inclusion visit or assessed no later than 8 days before randomization. To be eligible, the patient's electrolyte values should be within the following limits:

3.5 ≤ K+ ≤ 5 mmol/L 135 ≤ Na+ ≤ 145 mmol/L 2,20 ≤ Ca2+ ≤ 2,60 mmol/L

* Patient treated with a strong or moderate CYP3A4 inducer: carbamazepine, rifampicin, phenytoin, modafinil, efavirenz or a strong inhibitor of CYP3A4: azole antifungals, protease inhibitors, macrolids, without discontinuation ≥ 5 half-lives before randomization
* Patient treated with medicinal plants interacting with CYP3A4 without discontinuation ≥ 5 half-lives before randomization (Echinacea (E.pupurea, E.angustifolia and E.pallida), Piperina, Artemisia, St. John's Wort and Ginkgo Patient with Montreal Cognitive Assessment (MoCA) (Nasreddine et al., 2005) score < 20 (to exclude patients likely with dementia) at inclusion visit (Papay et al., 2014).
* Patient suffering from severe depression or marked suicidal thoughts (score > 3 on the suicidal thoughts item of the MADRS) at inclusion visit (Papay et al., 2014)
* History of DBS within the past year before randomization, or change in stimulation parameters less than one month prior to randomization Hematologic or solid malignancy diagnosis within 5 years prior to randomization.
* Patient suffering from severe renal impairment define as CrCL<30 mL/min, Cockcroft-Gault at inclusion visit or assessed no later than 8 days before randomization
* Clinically significant hepatic impairment
* Concurrent participation in another research involving a drug or medical device
* Patient with language barriers precluding adequate understanding or co-operation or who, in the opinion of the investigator, should not participate in the trial
* Treatment with an investigational treatment within 30 days prior to randomization
* Woman pregnant, nursing or of childbearing potential age without effective contraception methods or intends to become pregnant.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants randomized in the PIMPARK study (PHRC 2015-HUS 6398)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change in ICD (Impulsive Control Disorders) severity after 8 weeks of treatment evaluated by QUestionnaire for Impulse-compulsive disorder in Parkinson's disease Rating Scale (QUIP-RS). | at day 0 and week 8
  The primary endpoint of this study will be assessed in both arms using the total form of QUIP-RS.
  QUIP-RS has 4 primary questions (pertaining to commonly reported thoughts, urges/desires, and behaviors associated with ICDs), each applied to the 4 ICDs (compulsive gambling, buying, eating, and sexual behavior) and 3 related disorders (medication use, punding, and hobbyism). It uses a 5-point Likert scale (score 0-4 for each question) to gauge the frequency of behaviors. Scores for each ICD and related disorder range from 0 to 16 and the total QUIP-RS score for all ICDs and related disorders combined ranges from 0 to 112, with a higher score indicating greater severity (ie, frequency) of symptoms.

SECONDARY OUTCOMES:
Change SCale for Outcomes in Parkinson's disease - Sleep (SCOPA-SLEEP) score after 4 and 8 weeks of treatment | At day 0, week 4 and week 8
  The SCOPA-SLEEP is a specific Parkinson's disease rating scale for assessing nighttime sleep (NS) problems and daytime sleepiness (DS) in the past month. The NS subscale has 5 items, scored from 0 (not at all) to 3 (a lot). The DS subscale is composed of 6 items with response options ranging from 0 (never) to 3 (often) with a higher total score indicating greater severity of sleep problems.
Change SCale for Outcomes in Parkinson's disease - Sleep (Insomnia severity index) score after 4 and 8 weeks of treatment | At day 0, week 4 and week 8
  Scale ranging from 0 to 28 with a higher total score indicating greater severity of sleep problems.
Change SCale for Outcomes in Parkinson's disease - Sleep (PDSS-2: Parkinson Disease Sleep Scale-2) score after 4 and 8 weeks of treatment | At day 0, week 4 and week 8
  Scale ranging from 0 to 60 with a higher total score indicating greater severity of sleep problems.
Change in Movement Disorders Society-sponsored Unified Parkinson's Disease Rating scale (MDS-UPDRS) scores after 4 and 8 weeks of treatment | At day 0, week 4 and week 8
  MDS-UPDRS is a clinimetric assessment of subjective and objective symptoms and signs of Parkinson's disease. The MDS-UPDRS has four parts, namely, I: Non-motor Experiences of Daily Living; II: Motor Experiences of Daily Living; III: Motor Examination; IV: Motor Complications. The four parts contains 64 items which are each rated on a scale of 0 (normal or no disease effect) to 4 (maximum negative effect). Negative changes from baseline values indicate improvement
Change in Montgomery-Åsberg Depression Rating Scale (MADRS) scores after 4 and 8 weeks of treatment | At day 0, week 4 and week 8
  MADRS is a ten-item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders. Each item yields a score of 0 to 6 and the overall score ranges from 0 to 60 with higher MADRS score indicating more severe depression.
Change in Ardouin's scale scores after 4 and 8 weeks of treatment | At day 0, week 4 and week 8
  The Ardouin's scale is a validated instrument using a structured and standardised interview composed of 21 items specifically designed to assess mood and behaviour with a view to quantifying changes related to Parkinson's Disease, to dopaminergic medication, and to non-motor fluctuations. Each item is scored from 0 (absent) to 4 (severe).
Change in the rate of Clinical Global Impression Severity (CGIS) scale after 4, 8 and 16 weeks of treatment | At day 0, week 4, week 8 and week 16
  Severity of PD will be assessed in both arms using CGIS scale: the CGI-S is a 7-point scale that requires the rating of the severity of the patient's illness at the time of assessment. Possible ratings are: 1: Normal, not at all ill; 2: Borderline mentally ill; 3: Mildly ill; 4: Moderately ill ; 5: Markedly ill; 6: Severely ill; 7: Among the most extremely ill patients
Change in ICD (Impulsive Control Disorders) severity after 4 weeks of treatment evaluated by QUIP-RS. | At day 0 and week 4
  Global functioning and severity of the disease will be assessed in both arms by QUIP-RS has 4 primary questions each applied to the 4 ICDs and 3 related disorders It uses a 5-point Likert scale and a higher score indicating greater severity (ie, frequency) of symptoms.
Changes in quality of life measured by Parkinson's Disease Questionnaire (PDQ-39) scores after 4 and 8 weeks of treatment | At day 0, week 4 and week 8
  Functioning and well-being of patients during the preceding month will be assessed in both arms by 39 questions of the self-administered Parkinson's Disease Questionnaire (PQD-39). Each question is scored from 0 (never) to 4 (always), the higher score indicating higher impact of illness in quality of life.
Change in Zarit scale scores after 4 and 8 weeks of treatment for caregivers | At day 0, week 4 and week 8
  The burden of the patient's functional and behavioural worsening and to home care will be assessed to the caregiver in both arms by the Zarit Burden scale. It is composed of 22 items to measure the magnitude of the burden experienced by the caregiver. Each item is scored from 0 (never) to 4 (almost always). With a higher score indicating a greater load suffered by the caregiver.
Total number of adverse events and serious adverse events | At week 16
  Open-ended questionnaire will be used in both arms

CONTACTS AND LOCATIONS:
Locations (16):
- France (16):
  - Service de Neurologie et Centre d'Investigation Clinique CHRU de Besançon,, Besançon
  - SERVICE DE NEUROLOGIE Unité Mouvement anormaux Centre expert Parkinson (centre coordinateur interrégional pour la région Sud-Est) Service de neurologie C Hôpitaux Universitaires de Lyon Hôpital Neurologique Pierre Wertheimer, Bron
  - SERVICE DE NEUROLOGIE Unité Mouvement anormaux Centre expert Parkinson (région Sud-Est) Hôpitaux Universitaires de Clermont-Ferrand Hôpital Gabriel Montpied, Clermont-Ferrand
  - SERVICE DE NEUROLOGIE Pathologies du mouvement Centre expert Parkinson (région Ile-de-France) Hôpital Henri Mondor, Créteil
  - SERVICE DE NEUROLOGIE Pathologies du mouvement Centre expert Parkinson (région Sud-Est) CHU de Grenoble Alpes, Grenoble
  - SERVICE DE NEUROLOGIE Unité Mouvement anormaux Centre expert Parkinson (centre de coordination pour la région Nord-Ouest) Hôpitaux Universitaires de Lille Hôpital Roger Salengro, Lille
  - SERVICE DE NEUROLOGIE Pathologies du mouvement Centre expert Parkinson (région Sud-Ouest) Hôpitaux Universitaires de Limoges, Limoges
  - SERVICE DE NEUROLOGIE Unité Mouvement anormaux Centre expert Parkinson (centre de coordination pour la région Sud Méditerranée) Hôpitaux Universitaires de Marseille Hôpital La Timone, Marseille
  - SERVICE DE NEUROLOGIE Pathologies du mouvement Centre expert Parkinson (centre de coordination pour la région Ouest) Centre d'investigation clinique Hôpitaux Universitaires de Nantes, Nantes
  - SERVICE DE NEUROLOGIE Centre expert Parkinson (centre de coordination pour la région Ile-de-France) Hôpital de la Pitié-Salpêtrière, Paris
  - CIC Hôpitaux Universitaires de Poitiers, Poitiers
  - Service de neurologie, Hôpitaux Universitaires de REIMS, Reims
  - SERVICE DE NEUROLOGIE Pathologies du mouvement Centre expert Parkinson (région Ouest) Hôpitaux Universitaires de Rennes-Hôpital Pontchaillou, Rennes
  - SERVICE DE NEUROLOGIE Pathologies du mouvement Centre expert Parkinson (région Nord-Ouest) Hôpitaux Universitaires de Rouen Hôpital Charles Nicolle, Rouen
  - SERVICE DE NEUROLOGIE Unité Mouvement anormaux Centre expert Parkinson (centre de coordination pour la région Est) Hôpitaux Universitaires de Strasbourg Hôpital de Hautepierre, Strasbourg
  - SERVICE DE NEUROLOGIE Unité Mouvement anormaux Centre expert Parkinson/Centre d'Investigation Clinique -Hôpital Pierre-Paul Riquet, Toulouse

IPD SHARING:
Plan to Share IPD: No